CLINICAL TRIAL: NCT05770310
Title: A Phase I Study to Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of JS015 In Patients With Advanced Solid Tumors
Brief Title: A Phase I Study Of JS015 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS015-001-I
Record Dates: First submitted 2023-02-17; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Cancer

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS015 (Experimental)
  Interventions: Drug: JS015

INTERVENTIONS:
Drug: JS015 — Patient receives specific dose of JS015. The administration method of JS015 is intravenous infusion.

SUMMARY:
This is a Phase I open-label, multicenter study to evaluate the safety, tolerability, pharmacokinetics (PK), immunogenicity and antitumor activity of JS015 in patients with advanced solid tumors. The Recommended dose for phase II trial （RP2D） was determined based on the safety, pharmacokinetics, and initial efficacy data of the dose escalation and extension.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in this study and provide written informed consent;
2. Histologically- or cytologically-confirmed advanced solid tumors considered failure to the standard treatment, or with no standard treatment, or not available to standard treatment;
3. At least one measurable lesion according to RECIST 1.1;
4. Life expectancy ≥ 3 months;
5. Eastern Cooperative Oncology Group (ECOG) 0 or 1;
6. Adequate organ function;
7. Treatment related toxicities due to prior anti-cancer therapy including surgery and radiotherapy must be ≤ grade 1;
8. Women of childbearing age must confirm that the serum pregnancy test is negative within 7 days before the first dose; Male and female patients of child bearing potential will to use abstinence or an effective method of contraception throughout the treatment period and for 90 days following the last dose of study drug;

Exclusion Criteria:

1. Allergy or contraindication to JS015 and its ingredients;
2. Has a known additional malignancy in the last 5 years.
3. Pregnancy or lactation;
4. History of immunodeficiency, including human immunodeficiency virus(HIV) test positive, or known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
5. Brain or meningeal metastases
6. Pleural effusion, peritoneal effusion or pericardial effusion that required treatment (such as puncture, drainage)
7. Severe cardiovascular and cerebrovascular diseases;
8. Previous antineoplastic therapy meets washout requirements.
9. Severe infection (Criteria for the evaluation of common adverse events(CTC AE) 5.0>2 grade) occurred within 28 days before the first study administration; Active infection or unexplained fever > 38.5°C ;
10. Has active tuberculosis or hepatitis B (HBV) or hepatitis C (HCV);
11. moderate to severe that seriously affect lung function;
12. Other serious physical or mental diseases or laboratory abnormalities, or alcoholism, drug abuse, etc.,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
dose-limiting toxicity （DLT）、adverse event（AE）、serious adverse event（SAE） | 2Years
  incidence and severity of DLT, adverse events (AE), serious adverse events (SAE), Abnormal changes in laboratory and other tests with clinical significance
Maximum tolerated dose (MTD),RP2D | 2 Years
  Maximum tolerated dose (MTD), Recommended dose for phase II trial

SECONDARY OUTCOMES:
Peak concentration（Cmax） | 2 years
  The highest plasma drug concentration that can be achieved after medication
time to peak（Tmax） | 2 years
  After a single dose, the time of peak blood concentration
elimination half life（t1/2） | 2 years
  the time it takes the blood to reduce the concentration of the drug to half
immunogenicity | 2 years
  Incidence of Anti-Drug Antibody (ADA)
Objective response rate (ORR) based on Response Evaluation Criteria In Solid Tumors 1.1 (RECIST1.1) | 2 years
  Defined as the proportion of subjects who achieved partial response (PR) or complete response (CR)
overall survival (OS) | 2 years
  The time from randomization to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Medical Doctor, Principal Investigator — Affiliation: Shanghai Oriental Hospital; Jinming Yu, Medical Doctor, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (4):
- China (4):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai Oriental Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No